CLINICAL TRIAL: NCT04167618
Title: A Phase I/II Dose-escalation and Expansion Cohort Trial of Intracerebroventricular Radioimmunotherapy Using 177Lu-DTPA-Omburtamab in Pediatric and Adolescent Patients With Recurrent or Refractory Medulloblastoma
Brief Title: 177Lu-DTPA-Omburtamab Radioimmunotherapy for Recurrent or Refractory Medulloblastoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business priorities
Sponsor: Y-mAbs Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 301
Record Dates: First submitted 2019-11-11; First posted 2019-11-19 (Actual); Results first posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Medulloblastoma, Childhood
MeSH Terms: conditions — Medulloblastoma

STUDY DESIGN:
Intervention Model Description: Patients will receive up to two cycles in Part 1 and up to five cycles in Part 2 of intracerebroventricular 177Lu-DTPA-omburtamab. Safety and efficacy will be investigated during treatment and follow-up period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 177Lu-DTPA-omburtamab (Experimental): Intracerebroventricular administration of 177Lu-DTPA-omburtamab for up to two cycles (Part 1) and up to five cycles (Part 2).
  Interventions: Drug: 177Lu-DTPA-omburtamab

INTERVENTIONS:
Drug: 177Lu-DTPA-omburtamab — Biological, radiolabeled DPTA-omburtamab

SUMMARY:
Children and adolescents diagnosed with medullablastoma and with recurrent or refractory to frontline therapy will be treated with 177Lu-DTPA-omburtamab, which is a radioactive labelling of a murine monoclonal antibody targeting B7-H3.

DETAILED DESCRIPTION:
Part 1 is a dose-escalation phase with a 3+3 sequential-group design in which patients will receive a dosimetry dose followed by maximum of two 5-week cycles of treatment doses of intracerebroventricular 177Lu-DTPA-omburtamab.

Part 2 is a cohort-expansion phase in which patients will receive a maximum of five 5-week cycles of intracerebroventricular 177Lu-DTPA-omburtamab at the recommended dose determined in Part 1.

End of treatment will take place within 5 weeks after the last cycle and thereafter the patients will be enter the follow-up period. The patients will be followed for up to 2 years after last dose.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of medulloblastoma.
* SHH, Group 3, or Group 4 according to World Health Organisation (WHO) 2016 classification.
* Recurrent (maximum of 2 recurrences for Part 1 and 1 recurrence for Part 2) or refractory to frontline therapy. Prior frontline or second line therapy may involve surgery, craniospinal irradiation, stereotactic radiosurgery, and multi-agent chemotherapy regimens.
* Have refractory disease, focal or multifocal recurrent disease, or pure leptomeningeal disease. Cytological or radiographic remission is allowed; however, not simultaneously.
* Performance status score of 50 to 100 on Lansky (less than 16 years) or Karnofsky (16 years or older) scales.
* Life expectancy of at least 3 months, as judged by the Investigator.
* Acceptable hematological status and liver and kidney function.

Exclusion Criteria:

* Obstructive or symptomatic communicating hydrocephalus as determined by Ommaya patency/cerebrospinal fluid (CSF) flow study.
* Residual disease (nodular or linear) measuring > 15 mm in the smallest diameter.
* Ventriculoperitoneal shunts without programmable valves. Ventriculo-atrial or ventriculo-pleural shunts.
* Grade 4 nervous system disorder. Stable neurological deficits (due to brain tumor or surgery) or hearing loss are allowed.
* Uncontrolled life-threatening infection.
* Received radiation therapy less than 3 weeks prior to the screening visit.
* Received systemic or intrathecal cytotoxic chemotherapy or intrathecal immunotherapy (corticosteroids not included) less than 3 weeks prior to the screening visit.
* Received any prior anti-B7-H3 treatment.
* Non-hematologic organ toxicity Grade 3 or above; specifically, any renal, cardiac, hepatic, pulmonary, and gastrointestinal system toxicity.
* Other significant disease or condition that in the investigator's opinion would exclude the patient from the trial.

Ages: 3 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (4):
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Doernbecher Children's Hospital, Portland, Oregon
  - M.D. Anderson Cancer Center, Houston, Texas
- Rigshospitalet, Børneonkologisk afsnit, Copenhagen, Denmark
- Princess Máxima, Utrecht, Netherlands
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Sant Joan de Deu de Barcelona, Barcelona
- United Kingdom (2):
  - The Royal Marsden Hospital, London
  - Great North Children's Hospital, Newcastle

RESULTS

PARTICIPANT FLOW:
Groups:
- 10 mCi 177Lu-DTPA-omburtamab: Intracerebroventricular administration of 10 mCi 177Lu-DTPA-omburtamab for up to two cycles (Part 1).
  177Lu-DTPA-omburtamab: Biological, radiolabeled DPTA-omburtamab
- 25 mCi 177Lu-DTPA-omburtamab: Intracerebroventricular administration of 25 mCi 177Lu-DTPA-omburtamab for up to two cycles (Part 1).
  177Lu-DTPA-omburtamab: Biological, radiolabeled DPTA-omburtamab
Period: Overall Study
Arm/Group | 10 mCi 177Lu-DTPA-omburtamab | 25 mCi 177Lu-DTPA-omburtamab
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — Trial terminated by sponsor | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 mCi 177Lu-DTPA-omburtamab | 25 mCi 177Lu-DTPA-omburtamab | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 15 [15 to 15] | 8 [8 to 8] | 11.5 [8 to 15]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 0 | 1
  Denmark | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicities (DLTs) Part 1
Description: Summary of DLTs in DLT evaluable subjects.
Time Frame: Days 1 through 35 in cycle 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mCi 177Lu-DTPA-omburtamab | 25 mCi 177Lu-DTPA-omburtamab
Number analyzed (Participants) | 1 | 1
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: From 1st dose to 5 weeks after last dose, up to 10 weeks (2 cycles).
Arm/Group | 10 mCi 177Lu-DTPA-omburtamab | 25 mCi 177Lu-DTPA-omburtamab
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 mCi 177Lu-DTPA-omburtamab (N=1) | 25 mCi 177Lu-DTPA-omburtamab (N=1)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 mCi 177Lu-DTPA-omburtamab (N=1) | 25 mCi 177Lu-DTPA-omburtamab (N=1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood albumin decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial was terminated after 2 subjects due to a business strategy decision. At this point the maximum tolerated dose was not established.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-25): https://cdn.clinicaltrials.gov/large-docs/18/NCT04167618/Prot_SAP_000.pdf